CLINICAL TRIAL: NCT03917589
Title: Preventive Use of COrticosteroids During the Post-Partum in Relapsing MS
Brief Title: Preventive Use of COrticosteroids During the Post-Partum in Relapsing MS Patients (COPP-MS)
Acronym: COPP-MS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_9844_COPP-MS
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: post-partum; corticosteroids; relapse; disease modifying drugs (DMD)
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with corticosteroids: Patients who have systematically been treated by high-dose corticosteroids after the delivery
- Patients without corticosteroids: Patients who haven't been systematically treated by high-dose corticosteroids after the delivery.

SUMMARY:
Multiple Sclerosis (MS) is most prevalent among women of childbearing age. The post-partum (PP) period is a critical phase in MS patients, during which a recrudescence of disease activity is expected. Different strategies have been assessed in the prevention of post-partum relapse. High dose methylprednisolone was evaluated in a case control study with historical controls but the positive results have not been confirmed.

In this study, the main objective will be to compare the risk of relapse in the 6 months PP period between patients treated systematically by high dose methylprednisolone after delivery compared to patients who didn't receive a systematic treatment.

The second objective will be focused on the comparison of the disease activity and disability progression in patients who have resumed early a Disease Modifying Drug (DMD) after delivery vs patients who haven't.

DETAILED DESCRIPTION:
Even if two small case control studies underlined the positive effect of high dose methylprednisolone on the relapse risk in the PP period in MS, these data have to be confirmed by a larger study. The impact of such a strategy remains also uncertain concerning the risk of long term disability. In this project, the investigators will also analyze the influence of the delay of DMD reintroduction after delivery on the relapse risk but also on the risk of disability. The results will have an important role in the therapeutic management of the post-partum period in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing MS patients according to MacDonald criteria 2010
* Age between 15 and 49 years old at the pregnancy
* Age between 18 and 51 years old when filling the questionnaire of the study
* At least one full pregnancy with live birth after the beginning of the MS diagnosis
* At least one neurological visit during the 12 months period after the delivery
* At least one neurological visit per year in the 12 months preceding the pregnancy
* Pregnancy must occur between 01/2007 and 01/2017 In case of several pregnancies per woman, only the first one occurring in the period will be analyzed
* Having received information on the protocol and not having expressed opposition to participating in the study.

Exclusion Criteria:

* Patients who have received Immunoglobulines or plasma exchanges after the delivery in prevention of a relapse
* Patients presenting a SPMS or PPMS form at the beginning of pregnancy
* Protected persons referred to in Articles L. 1121-6 to L. 1121-9 of the code of public health (eg minors, persons deprived of liberty, ..) except nursing mothers postpartum.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Study of Preventive use of COrticosteroids during the Post-Partum
Study Population: relapsing MS patients with at least one full pregnancy with live birth between 01/2007 and 01/2017 after the beginning of the MS diagnosis
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Difference of the proportion of patients with >= 1 relapse between the two groups | 6 months
  proportion of patients with >= 1 relapse during the six-month period after delivery between the patients who have systematically been treated by high-dose corticosteroids after the delivery; and patients who haven't been systematically treated by high-dose corticosteroids.

SECONDARY OUTCOMES:
Difference of the proportion of patients with >= 1 relapse | 6 months
  proportion of patients with >= 1 relapse during the six-month period after delivery between patients who have resumed a DMD early after the delivery (during the first two months) compared to a delayed reintroduction, or an absence of reintroduction
Difference of the annualized relapse rate | 6 months
  Number of the annualized relapse rate after the delivery between corticosteroids or not and between early DMD vs delayed DMD
Difference of the annualized relapse rate | 1 year
  Number of the annualized relapse rate after the delivery between corticosteroids or not and between early DMD vs delayed DMD
Difference of the annualized relapse rate | two years
  Number of the annualized relapse rate after the delivery between corticosteroids or not and between early DMD vs delayed DMD
Difference of the time to first relapse | Date of delivery
  Time to first relapse after delivery between corticosteroids or not and between early DMD vs delayed DMD
Difference of the disability progression | 6 months
  Score of Expanded Disability Status Scale (EDSS) (from 0=no disability, to 10= Death / No sub scales) between corticosteroids or not and between early DMD vs delayed DMD
Difference of the disability progression | 1 year
  Score of Expanded Disability Status Scale (EDSS) (from 0=no disability, to 10= Death / No sub scales) between corticosteroids or not and between early DMD vs delayed DMD
Difference of the disability progression | 2 years
  Score of Expanded Disability Status Scale (EDSS) (from 0=no disability, to 10= Death / No sub scales) between corticosteroids or not and between early DMD vs delayed DMD
Difference of percentage of with Gadolinium enhancing lesions | 6 months
  Difference of percentage of with Gadolinium enhancing lesions during the 6-month period after the delivery between corticosteroids or not and between early DMD vs delayed DMD
Difference of the number of Gadolinium enhancing lesions | 6 months
  compare the number of Gadolinium enhancing lesions during the 6-month period after the delivery between corticosteroids or not and between early DMD vs delayed DMD

CONTACTS AND LOCATIONS:
Overall Officials: Laure MICHEL, Dr, Principal Investigator — CHU Rennes
Locations (5):
- France (5):
  - Hôpital LAENNEC, Saint-Herblain, Nantes
  - CHU Lyon, Lyon
  - Hôpital Pasteur 2 - CHU Nice, Nice
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No